CLINICAL TRIAL: NCT05440422
Title: The Role of Anifrolumab in Improving Markers of Vascular Risk in Patients With Systemic Lupus Erythematosus
Brief Title: The Role of Anifrolumab in Improving Markers of Vascular Risk in Patients With Systemic Lupus Erythematosus (SLE) - IFN-CVD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 10000682; 000682-AR
Record Dates: First submitted 2022-06-29; First posted 2022-06-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Systemic Lupus Erythematosus; Cardiovascular Disease; Premature Atherosclerosis
Keywords: Vascular Inflammation; Interferons; Vascular Function
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Cardiovascular Diseases | interventions — anifrolumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patient (Active Comparator): anifrolumab
  Interventions: Drug: anifrolumab
- Patient placebo (Placebo Comparator): placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: anifrolumab — This is a double blind placebo-controlled study to characterize whether blocking type I IFN receptor signaling with anifrolumab will lead to improvements in vascular function, decreases in vascular inflammation and modulation of biomarkers of vascular risk in patients with SLE.
  Arms: Patient
Other: Placebo — non-active substance comprised of 25 mM histidine/histidine-HCl, 50 mM lysine-HCl, 130 mM trehalose, and 0.05% (w/v) polysorbate 80, with a pH of 5.9.
  Arms: Patient placebo

SUMMARY:
Background:

People with systemic lupus erythematosus (SLE) are at risk of developing complications in their blood vessels. This can increase the risk of heart attacks or stroke. No medications have been effective at reducing this risk in people with lupus.

Objective:

To test whether a drug (anifrolumab) can improve blood vessel function and reduce blood vessel inflammation in people with SLE.

Eligibility:

People aged 18 to 80 years with SLE.

Design:

Participants will undergo screening. They will have a physical exam. They will have blood and urine tests. They will have a test of their heart function and a chest X-ray. They will answer questions about their SLE symptoms.

Participants will visit the clinic 9 times in 8 months. After screening, visits will be 4 weeks apart. Each visit may take up to 4 hours.

Participants will receive infusions from a tube attached to a needle inserted into a vein in the arm (IV). Some will receive anifrolumab. Others will receive a placebo treatment. They will not know which one they are getting.

At some visits they will have additional tests:

CAVI (cardio-ankle vascular index) tests blood vessel function. Participants will lie still for 20 minutes. Small electrodes will be placed on both wrists with stickers. A microphone will be placed on their chest. Blood pressure cuffs will be wrapped around their ankles and arms.

FDG-PET/CT is an imaging procedure. Participants will receive a substance through an IV line. They will lie on a table for 110 minutes while a machine captures images of their body.

DETAILED DESCRIPTION:
Study Description:

This is a double blind placebo-controlled study to characterize whether blocking type I IFN receptor signaling with anifrolumab will lead to improvements in vascular function, decreases in vascular inflammation and modulation of biomarkers of vascular risk in patients with systemic lupus erythematosus (SLE).

Objectives:

Primary Objective:

To assess the role of anifrolumab in modulating vascular function and vascular inflammation in SLE patients with mild to moderate disease activity as determined by Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) 2K<= 6.

Secondary Objectives:

To assess the role of anifrolumab in modulating biomarkers of cardiovascular risk in SLE patients with mild to moderate disease activity as determined by SLEDAI 2K<= 6. Assess safety and tolerability of short-term use of anifrolumab

Endpoints:

Primary:

1. Change from Baseline (Week 0) to Week 28 in cardio-ankle vascular index (CAVI).
2. Change from Baseline to Week 28 in pulse wave velocity (PWV) using Sphygmocor.
3. Change from Baseline to Week 28 in vascular inflammation as measured by target to background ratio (TBR) in various aortic territories and total aorta using FDG PET CT scans.

Secondary:

Changes over time in biomarkers of cardiovascular risk/immune dysregulation and metabolic dysfunction previously described in SLE. These biomarkers include but not limited to lipoprotein profiles and high-density lipoprotein cholesterol efflux capacity, immune cell types, endothelial progenitor cells, circulating neutrophil extracellular traps, serum cytokines, acute phase reactants, insulin resistance, transcriptomic analysis of peripheral immune cells.

Tertiary:

Safety, as assessed by severity and incidence of adverse events and the change over time from baseline in laboratory variables.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18-80 years
4. In good general health as evidenced by medical history or diagnosed with SLE diagnosed per American College of Rheumatology 1997 revised SLE classification criteria.
5. Prednisone < or equal to 10 mg/day for at least 2 weeks before screening and maintained throughout randomization (day 1)
6. Stable standard of care lupus therapies for at least 4 weeks before screening and maintained through randomization (day 1)
7. Abnormal cardio-ankle vascular index(CAVI) at screening OR up to 90 days prior to the screening visit (based on 2 SD above median of healthy controls based on historical data from our own patient cohorts
8. Stable medications for diabetes, hypertension and/or statins for at least the previous 3 months. No changes of these medications or immunosuppressive drugs will be allowed during trial.
9. For females and males of reproductive potential: use of highly effective contraception from screening and agreement to use such a method during study participation and for an additional 16 weeks after the end of study medication administration. For the purpose of this study abstinence will be considered as an effective form of contraception.
10. Subjects must confirm receipt of prior vaccination against COVID-19 and Varicella Zoster. Verbal confirmation of vaccination receipt AND detectable antibodies in serum is acceptable in the absence of vaccine records.

    EXCLUSION CRITERIA:

    An individual who meets any of the following criteria will be excluded from participation in this

    study:
    * Any condition that, in the opinion of the Investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.
    * Concurrent enrolment in another clinical study with an investigational product
    * Major surgery within 8 weeks before signing the ICF or elective major surgery planned during the study period.
    * Any of the following found at Screening:

      * Aspartate aminotransferase (AST) >2.5 x upper limit of normal (ULN).
      * Alanine aminotransferase (ALT) >2.0 x ULN.
      * Total bilirubin >ULN (unless due to Gilbert's syndrome)
      * Serum creatinine >2.5 mg/dL (or >181 micromol/L)
      * Urine protein/creatinine ratio >2.0 mg/mg (or >226.30 mg/mmol)
      * Neutrophil count <1000/microL (or <1.0 x 109/L)
      * Platelet count <25000/microL (or <25 x 109/L)
      * Hemoglobin <8 g/dL (or <80 g/L), or <7 g/dL (or <70 g/L) if related to subject's SLE such as in active hemolytic anemia
      * Glycosylated hemoglobin (HbA1c) >8% (or >0.08) at screening (diabetic subjects only)
      * Positive SARS/Flu A/B/RSV (Panther), PCR

    Note: Abnormal screening test(s) which exclude the patient may be repeated once within 4 weeks of the Screening Visit. If the repeat test(s) does not meet the above criteria, then the patient may be included in the study and will not be considered a screen failure.
    * Receipt of any of the following:

      1. Azathioprine >200 mg/day
      2. Mycophenolate mofetil > 3 g/day or mycophenolic acid >2.16 g/day
      3. Oral, SC, or intramuscular methotrexate >25 mg/week
      4. Mizoribine >150 mg/day. Leflunomide more than 20 mg and any other immunosuppressant usage at the discretion of the PI.
    * Receipt of any investigational product (small molecule or biologic agent) within 4 weeks or 5 half-lives prior to week 0 (day 1), whichever is greater.
    * Receipt of any commercially available biologic agent within 5 half-lives prior to signing of the ICF
    * Receipt of B cell depleting therapy (including but not limited to belimumab, ocrelizumab, ofatumumab, atacicept, Obinutuzumab, or rituximab), <26 weeks prior to the signing of the consent for all B-cell depleting therapy or <40 weeks prior to the signing of the ICF for atacicept.
    * Receipt of any of the following: (a) Intra-articular, intramuscular or IV corticosteroids within 4 weeks prior to Day 1 (b) Any live or attenuated vaccine within 8 weeks prior to signing the ICF (administration of killed vaccines is acceptable)
    * History or evidence of suicidal ideation within the past 6 months; or any suicidal behavior within the past 12 months based on screening or at baseline.
    * Recent cardiac or stroke event (with in the last year prior to week 0 (day 1))
    * Active SLE disease with SLEDAI 2K >6 at the time of screening.
    * Active severe or unstable neuropsychiatric SLE including, but not limited to: aseptic meningitis; cerebral vasculitis; myelopathy; demyelination syndromes (ascending, transverse, acute inflammatory demyelinating polyradiculopathy); acute confusional state; impaired level of consciousness; psychosis; acute stroke or stroke syndrome; cranial neuropathy; status epilepticus; cerebellar ataxia; and mononeuritis multiplex:

      1. That would make the subject unable to fully understand the ICF OR
      2. Where, in the opinion of the Principal Investigator (PI), protocol specified SOC is insufficient and utilization of a more aggressive therapeutic approach, such as adding IV cyclophosphamide and/or high dose IV pulse corticosteroid therapy or other treatments not permitted in the protocol, is indicated
    * Active severe SLE-driven renal disease where, in the opinion of the PI, protocol specified standard of care (SOC) is insufficient and utilization of a more aggressive therapeutic approach, such as adding IV cyclophosphamide and/or high dose IV pulse corticosteroid therapy or other treatments not permitted in the protocol, is indicated.
    * History of or current diagnosis of catastrophic or severe anti-phospholipid syndrome within 1 year prior to signing the ICF. Antiphospholipid syndrome adequately controlled by anticoagulant therapy for at least 3 months is acceptable.
    * Known history of a primary immunodeficiency, splenectomy, or any underlying condition that predisposes the subject to infection, or a positive result for human immunodeficiency virus (HIV) infection confirmed by central laboratory at screening. Subjects refusing HIV testing during the screening period will not be eligible for study participation.
    * Confirmed positive test for hepatitis B serology for:

      1. Hepatitis B surface antigen (HBsAg), OR
      2. Hepatitis B core antibody (HBcAb)
      3. If positive for HBcAb, hepatitis B virus (HBV) DNA will be checked. If HBV DNA is detected above the lower limit of quantitation (LLOQ) at screening subject will be excluded

    Note: Subjects who are only HBcAb positive at screening will be tested every month for HBV DNA. To remain eligible for the study, the subject s HBV DNA levels must remain below the LLOQ as per the central laboratory.
    * Positive test for hepatitis C antibody along with detectable Hepatitis C viral RNA.
    * Any severe herpes infection at any time prior to Week 0 (Day 1), including, but not limited to, disseminated herpes (ever), herpes encephalitis (ever), recurrent herpes zoster (defined as 2 episodes within 2 years) or ophthalmic herpes (ever)
    * Any herpes zoster, cytomegalovirus (CMV) or Epstein-Barr virus infection that has not completely resolved within 12 weeks prior to signing the ICF.
    * Any of the following:

      1. Clinically significant chronic infection (i.e., osteomyelitis, bronchiectasis, etc.) within 8 weeks prior to week 0 (day1) (chronic nail infections are allowed)
      2. Any infection requiring hospitalization or treatment with IV antibiotics not completed at least 4 weeks prior to week 0 (day1)
    * Any infection requiring oral antimicrobials (including antivirals) within 2 weeks prior to Day 1, except if taking antivirals/antimicrobials prophylactically.
    * History of cancer, apart from:

      1. Squamous or basal cell carcinoma of the skin treated with documented success of curative therapy >=3 months prior to Week 0 (Day 1)
      2. Cervical cancer in situ treated with apparent success with curative therapy >=1 year prior to Week 0 (Day 1).
    * Pregnancy or lactation or intend to become pregnant anytime from initiation of Screening until completion of study.
    * Spontaneous or induced abortion, still or live birth, or pregnancy <= 4 weeks prior to week 0 (day1)
    * Known allergic reactions to any component of the investigational product formulation or history of anaphylaxis to any human gamma globulin therapy.
    * Tested positive for COVID-19 infection on the day of screening or up to 21 days prior to screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-02 (Estimated)

PRIMARY OUTCOMES:
role of anifrolumab | 8 months
  1.Change from Baseline (Week 0) to Week 28 in cardio-ankle vascular index (CAVI). 2. Change from Baseline to Week 28 in pulse wave velocity (PWV) using Sphygmocor. 3. Change from Baseline to Week 28 in vascular inflammation as measured by target to background ratio (TBR) in various aortic territories and total aorta using FDG PET CT scans.

SECONDARY OUTCOMES:
Role of anifrolumab | 8 months
  in modulating biomarkers of cardiovascular risk in SLE patients with mild to moderate disease activity as determined by SLEDAI 2K= 6. Assess safety and tolerability of short-term use of anifrolumab

CONTACTS AND LOCATIONS:
Overall Officials: Mariana J Kaplan, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
The protocol is silent on sharing IPD.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000682-AR.html